CLINICAL TRIAL: NCT04761978
Title: Effectiveness and Safety of JAK Inhibitors for the Treatment of Moderate-to-severe Atopic Dermatitis in a Real-life French Multicenter Adult Cohort
Brief Title: Efficacy and Tolerance of JAK Inhibitors in ATU for Atopic Dermatitis
Acronym: JAKIGREAT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: NI_2021_01
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Dermatitis, Atopic
Keywords: Effectiveness; Safety; JAK inhibitors; Atopic dermatitis; Adults
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is to assess effectiveness (EASI, SCORAD, IGA, DLQI, pruritus, sleep loss) and safety (clinical and biological adverse events) of JAK inhibitors in adults with moderate-to-severe atopic dermatitis in a real-life French multicenter retrospective cohort

ELIGIBILITY:
Inclusion Criteria:

* Adults
* moderate to severe atopic dermatitis
* treated by JAK inhibitors between december 2020 and september 2021
* inefficiency, loss of efficiency or contra-indication of previous systemic agent, DUPILUMAB or phototherapy
* ineligibility to French ongoing clinical trials

Exclusion Criteria:

* Children
* mild atopic dermatitis
* eligibility to CICLOSPORINE, METHOTREXATE, DUPILUMAB, phototherapy
* eligibility to French ongoing clinical trials
* patients' opposition for the use of their records
* follow up <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients assessed by French members of the Groupe de Recherche sur l'Eczema Atopique.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
reduction in Eczema Area and Severity Index (EASI) | At 3 months

SECONDARY OUTCOMES:
SCORing Atopic Dermatitis (SCORAD) | at baseline and at 3 months
Investigator's Global Assessment (IGA) | at baseline and at 3 months
Dermatology Life Quality Index (DLQI) | at baseline and at 3 months
patient-reported pruritus score from 0 to 10 | at baseline and at 3 months
patient-reported sleep loss from 0 to 10 | at baseline and at 3 months
Adverse effects (biological and clinical) | at baseline and at 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Staumont-Salle, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lisle-sur-Tarn, France